CLINICAL TRIAL: NCT01330550
Title: Effect of High Fiber and Sugar Free Biscuits in Diabetics Population
Brief Title: Effect of High Fiber and Sugar Free Biscuits in Prediabetics Population
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Hui-Ying, Huang/associate professor, China Medical University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: DMR99-IRB-209
Record Dates: First submitted 2011-03-09; First posted 2011-04-07 (Estimated); Last update posted 2011-04-07 (Estimated); Status verified 2011-04

CONDITIONS: Impaired Glucose Tolerance
Keywords: High fiber sugar free biscuit; pre-diabetics
MeSH Terms: conditions — Glucose Intolerance

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- high fiber sugar free biscuit. (Experimental): High fiber sugar free biscuit will regulate Blood sugars.
  Interventions: Dietary Supplement: High fiber sugar free biscuit

INTERVENTIONS:
Dietary Supplement: High fiber sugar free biscuit — Dosage form:Biscuit, Dosage:1.94gram fiber/slice, Frequency:9 slices/meal;3 times/day. Duration:8 weeks
  Other Names: Taiwan IMeI high fiber sugar free biscuit

SUMMARY:
The increase in diabetic population of the world is among the top ten causes of death; with diabetes always high on the list of causes of death. Diabetes is always relative to other major causes of death, (e.g. in cerebral vascular disease, cardiovascular disease and renal disease).

The eating habits and patterns of the diabetic patient are the main causes for poor glycemic control. In epidemiological studies, high fiber and low sugar dietary intake can significantly reduce the incidence of diabetes.

The purpose of this study is to investigate the effect of high fiber sugar-free biscuits in regulating blood glucose in pre-diabetic subjects.

The study will be conducted in three periods:

Period-I:

The recruitment of 60 pre-diabetic subjects:

Subjects of blood glucose levels "Impaired fasting glucose; IFG": fasting blood glucose ≧ 100 mg / dL, < 126 mg / dL or "Impaired glucose tolerance; IGT": 2 hours postprandial blood glucose ≧ 140mg/dL, < 200 mg/dL or clinically judged to be mild or moderate diabetes mellitus (HbA1c < 9%).

In addition to perform pre-test, all subjects also need to complete nutrition counseling and nutrition education .

All 60 subjects are randomly selected into two groups, Group-1,30 subjects, (Placebo group, normal fiber and normal sugar biscuit group), Group-2, 30 subjects, (Experimental group, high fiber and sugar free biscuit group)

The period-II:

Duration: 8 weeks Group-1,30 subjects, (Placebo group, normal fiber and normal sugar biscuit group) , All 30 subjects consume 3 servings of Low-fiber, normal sugar biscuits daily.

Group-2, 30 subjects, (Experimental group, high fiber and sugar free biscuit group) All 30 subjects consume 3 serving of high-fiber, and sugar free biscuits (containing 16 grams of fiber) daily.

Post-period:

Blood samples of all 60 subjects will be collected to compare with period-I and period-II at the first day of 9th week.

Report of expectation:

The purpose of this study is to help the pre-diabetic subjects to reduce the risk of becoming diabetic through the consuming of high fiber and sugar free biscuits and nutrition education.

DETAILED DESCRIPTION:
The increase in diabetic population of the world, is among the top ten causes of death; with diabetes always a top cause of death. Diabetes is always related with other major causes of death, (e.g. in cerebral vascular disease, cardiovascular disease and renal disease).

The eating habits and patterns of diabetic patient are the main causes for poor glycemic control. In epidemiological studies, high fiber rand low sugar dietary intake can significantly reduce the incidence of diabetes.

The purpose of this study is to investigate the effect of high fiber sugar-free biscuits in regulating blood glucose in pre-diabetic subjects.

The study will be conducted in three periods:

Period-I:

The recruitment of 60 pre-diabetic subjects:

Subjects of blood glucose levels "Impaired fasting glucose; IFG": fasting blood glucose ≧ 100 mg / dL, < 126 mg/dL or "Impaired glucose tolerance; IGT": 2 hours postprandial blood glucose ≧ 140mg/dL, < 200 mg/dL or clinically judged to be mild or moderate diabetes mellitus (HbA1c < 9%) .

In addition to perform pre-test, all subjects also need to complete nutrition counseling and nutrition education .

All 60 subjects are randomly selected into two groups, Group-1,30 subjects, (Placebo group, normal fiber and normal sugar biscuit group) , Group-2, 30 subjects, (Experimental group, high fiber and sugar free biscuit group)

Blood samples will be collected from all 60 subjects to investigate:

HbA1c, Blood sugars(Fasting and 2 hours after meal), Insulin, Fructosamine, SGOT,SGPT,ALK-P,TOTAL PROTEIN, Albumin, Globulin, Ketone, Bun,Creatinine, Cholesterol,TG,LDl,HDL, WBC,RBC,Hgb,Hct,M.C.V.,MCH,MCHC,Platelet.

The period-II:

Duration: 8 weeks Group-1,30 subjects, (Placebo group, normal fiber and normal sugar biscuit group), All 30 subjects consume 3 serving of Low-fiber, normal sugar biscuits daily.

Group-2, 30 subjects,(Experimental group, high fiber and sugar free biscuit group) All 30 subjects consume 3 serving of high-fiber, and sugar free biscuits(containing 16 grams of fiber) daily.

Post-period:

Blood samples of all 60 subjects will be collected to compare with period-I and period-II at the first day of 9th week.

Report of expectation:

The purpose of this study is to help the pre-diabetic subjects to reduce the risk of becoming diabetic through the consuming of high fiber and sugar free biscuits and nutrition education.

ELIGIBILITY:
Inclusion Criteria:

* fasting blood glucose ≧100mg/dL and < 126mg/dL
* Impaired glucose tolerance; IGT
* HbA1c < 9%

Exclusion Criteria:

* DM patients
* Pregnant

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-03; Primary Completion 2011-10 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
HbA1c | up to 8 weeks
  The investigators expect the HbA1c will be greatly improved at the end of the study.

SECONDARY OUTCOMES:
Insulin, Fasting Glucose,Ketone Body, Fructosamine. | 8 weeks
  The investigators expect the following data will be improved at the end of the study:Insulin, Fasting Glucose, Ketone Body, Fructosamine.

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University, Taichung, Taiwan